CLINICAL TRIAL: NCT03318471
Title: The Effect of Intravenous Single Dose of Magnesium Sulphate on Attenuation of Hemodynamic Pressor Response After Myfield's Clamp Application During Craniotomies
Brief Title: Magnesium Sulphate for Attenuation of Hemodynamic Pressor Response After Myfield's Clamp Application
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: El-Sahel Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Samir Ahmed Ahmed ElKafrawy, Fellow of Anesthesia & Pain Relief, El-Sahel Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017101
Record Dates: First submitted 2017-10-14; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Supratentorial Brain Tumor
Keywords: MgSo4, Mayfield clamp, pressor effect
MeSH Terms: interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Active Comparator): received 50 mg/kg MgSo4 in 100 ml 0.9 NaCl 15 minutes prior to anesthesia induction over 15 minutes
  Interventions: Drug: MgSo4
- Group S (Placebo Comparator): received 100 ml 0.9% NaCl 15 minutes prior to anesthesia induction over 15 minutes.
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: MgSo4 — 50 mg/kg MgSo4 in 100 ml 0.9 sodium Chloride 15 minutes prior to anesthesia induction over 15 minutes
  Other Names: magnesium sulphate
  Arms: Group M
Drug: 0.9% NaCl — 100 ml 0.9% NaCl 15 minutes prior to anesthesia induction over 15 minutes
  Other Names: normal saline
  Arms: Group S

SUMMARY:
Use of Mayfield skull clamp during craniotomies; results in a sharp and intense noxious stimulus which results in a severe hemodynamic pressor response. Many strategies have been reported to blunt this undesirable pressor effect. This prospective, double blind, and randomized study is the first to evaluate the effect of MgSo4 on attenuation of hemodynamic pressor activity after head clamp application during craniotomies.

DETAILED DESCRIPTION:
Background: Use of Mayfield skull clamp during craniotomies; results in a sharp and intense noxious stimulus which results in a severe hemodynamic pressor response. Many strategies have been reported to blunt this undesirable pressor effect. This prospective, double blind, and randomized study is the first to evaluate the effect of MgSo4 on attenuation of hemodynamic pressor activity after head clamp application during craniotomies.

Methods: This randomized, double blind, and prospective study was done in Neurosurgical department at ElSahel Teaching Hospital in Cairo from February 2016 till august 2017. All adult patients aged from 18 to 60 years of both genders, ASA physical status I and II scheduled for craniotomies were assessed to enter this study. Seventy one patients were assessed preoperatively, sixty of them were enrolled and assigned in two groups (n=30 each). Group M received 50 mg/kg MgSo4 in 100 ml 0.9 sodium Chloride 15 minutes prior to anesthesia induction over 15 minutes. Group S received 100ml 0.9% Sodium Chloride over the same period with the same rate.Mean HR was recorded as a primary outcome , meanwhile; MAP and the need for a bolus dose of fentanyl was considered a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged from 18 to 60 years
* of both genders
* ASA physical status I and II
* scheduled for craniotomies

Exclusion Criteria:

* history of MgSo4 consumption or allergy
* renal disease
* hepatic or endocrine disorder
* cardiovascular dysfunction
* calcium channel blocker intake
* drug abuse were excluded from this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Mean HR | From time of insertion over 30 minutes period {at the time of pins insertion (Pin 0),60 seconds ( pin 60'), 5 minutes (pin 5''), 10 minutes ( pin 10''), 20 minutes ( pin 20'') and 30 minutes (pin 30'').}
  Mean heart rate/min.

SECONDARY OUTCOMES:
MAP | From time of insertion over 30 minutes period {at the time of pins insertion (Pin 0),60 seconds ( pin 60'), 5 minutes (pin 5''), 10 minutes ( pin 10''), 20 minutes ( pin 20'') and 30 minutes (pin 30'').}
  Mean arterial Blood Pressure (mmHg)
Need for a bolus opioid | from time of insertion over 30 minutes .
  Need for a bolus fentanyl after pins insertion to alleviate pressor effects

CONTACTS AND LOCATIONS:
Overall Officials: Samir A ElKafrawy, MD, Principal Investigator — ElSahel Teaching hospital,Cairo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Gonzales RM, Masone RJ, Peterson R. Hemodynamic response to application of neurosurgical skull-pin head-holder. Anesth Rev. 1987; 14:53-4.
- [Background] Bithal PK, Dash HH, Chauhan R, Mohanty B. Haemodynamic changes in response to skull-pins application - Comparison between normotensive and hypertensive patients. Indian J Anaesth. 2002; 46:383-5.
- [Background] Paul A, Krishna HM. Comparison between intravenous dexmedetomidine and local lignocaine infiltration to attenuate the haemodynamic response to skull pin head holder application during craniotomy. Indian J Anaesth. 2015 Dec;59(12):785-8. doi: 10.4103/0019-5049.171558. PMID 26903671
- [Background] Osborn I, Sebeo J. "Scalp block" during craniotomy: a classic technique revisited. J Neurosurg Anesthesiol. 2010 Jul;22(3):187-94. doi: 10.1097/ANA.0b013e3181d48846. PMID 20479675